CLINICAL TRIAL: NCT01990612
Title: Induction in Nulliparous Women at 39 Weeks to Prevent Adverse Outcomes: A Randomized Controlled Trial
Brief Title: A Randomized Trial of Induction Versus Expectant Management
Acronym: ARRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD36801-ARRIVE; UG1HD027869 (NIH); UG1HD027915 (NIH); UG1HD034116 (NIH); UG1HD034208 (NIH); UG1HD040500 (NIH); UG1HD040485 (NIH); UG1HD040544 (NIH); UG1HD053097 (NIH); UG1HD040545 (NIH); UG1HD040560 (NIH); UG1HD087230 (NIH); UG1HD087192 (NIH); UG1HD040512 (NIH); UG1HD068258 (NIH); UG1HD068268 (NIH); U10HD036801 (NIH); UG1HD068282 (NIH)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Labor and Delivery
Keywords: Induction of labor; Expectant management of labor; 39 weeks gestation

STUDY DESIGN:
Intervention Model Description: Randomized trial of 6000 women at 38 weeks 0 days to 38 weeks 6 days randomized to one of two arms: elective induction of labor between 39 weeks 0 days and 39 weeks 4 days; or expectant management (unless a medical indication arises) until at least 40 weeks 5 days.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expectant Management (No Intervention): Expectant management (unless a medical indication arises) until at least 40 weeks 5 days.
- Elective Induction of Labor (Other): Elective induction of labor between 39 weeks 0 days and 39 weeks 4 days
  Interventions: Procedure: Elective Induction of Labor

INTERVENTIONS:
Procedure: Elective Induction of Labor — Women randomized to induction of labor will undergo induction via oxytocin at 39 weeks 0 days to 39 weeks 4 days. Those with an unfavorable cervix (modified Bishop score < 5) will first undergo cervical ripening (method left to the discretion of the patient's physician) in conjunction with or followed by oxytocin stimulation unless a contraindication arises.
  Arms: Elective Induction of Labor

SUMMARY:
A randomized clinical trial to assess whether elective induction of labor at 39 weeks of gestation compared with expectant management will improve outcomes.

DETAILED DESCRIPTION:
Given the reported increased risks of adverse events in pregnancies extending beyond 39 weeks it has been hypothesized that a policy of planned elective induction at 39 weeks could improve outcomes for the infant and the mother. For multiparous patients, especially those with a favorable cervix, it is perhaps easy to justify an elective induction at 39 weeks given the low risk of cesarean section. However, for nulliparous patients the current evidence, derived mainly from retrospective observational studies, does not allow a clear recommendation. Nevertheless, a trend towards an increased rate of elective labor induction in pregnancies at 39 weeks has been reported, indicating that practitioners are more commonly using elective induction at this gestational age,even as others caution against routine elective induction prior to 41 weeks given the reported increased risk of cesarean delivery. Ultimately, a randomized controlled trial is necessary to satisfactorily understand whether elective induction of labor of nulliparas at 39 weeks improves neonatal and maternal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous - no previous pregnancy beyond 20 weeks
2. Singleton gestation. Twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks project gestational age.
3. Gestational age at randomization between 38 weeks 0 days and 38 weeks 6 days inclusive based on clinical information and evaluation of the earliest ultrasound.

Exclusion Criteria:

1. Project gestational age at date of first ultrasound is > 20 weeks 6 days
2. Plan for induction of labor prior to 40 weeks 5 days
3. Plan for cesarean delivery or contraindication to labor
4. Breech presentation
5. Signs of labor (regular painful contractions with cervical change)
6. Fetal demise or known major fetal anomaly
7. Heparin or low-molecular weight heparin during the current pregnancy
8. Placenta previa, accreta, vasa previa
9. Active vaginal bleeding greater than bloody show
10. Ruptured membranes
11. Cerclage in current pregnancy
12. Known oligohydramnios, defined as AFI < 5 or MVP < 2
13. Fetal growth restriction, defined as EFW < 10th percentile
14. Known HIV positivity because of modified delivery plan
15. Major maternal medical illness associated with increased risk for adverse pregnancy outcome (for example, any diabetes mellitus, lupus, any hypertensive disorder, cardiac disease, renal insufficiency)
16. Refusal of blood products
17. Participation in another interventional study that influences management of labor at delivery or perinatal morbidity or mortality
18. Delivery planned elsewhere at a non-Network site

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6106 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Miodovnik, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Rebecca Clifton, PhD, Principal Investigator — The George Washington University Biostatistics Center; William Grobman, MD, Study Chair — Northwestern University
Locations (16):
- United States (16):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Colorado
  - Northwestern University-Prentice Hospital, Chicago, Illinois
  - Columbia University-St. Luke's Hospital, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Dept of OB/GYN, Southwestern Medical Center, University of Texas, Dallas, Texas
  - University of Texas - Galveston, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses. Requests for datasets can be sent to mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Result] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Derived] Mallett G, Hill K, Doherty L, Grobman WA, Reddy UM, Tita ATN, Silver RM, Rice MM, El-Sayed YY, Wapner RJ, Rouse DJ, Saade GR, Thorp JM Jr, Chauhan SP, Costantine MM, Chien EK, Casey BM, Srinivas SK, Swamy GK, Simhan HN, Macones GA; The Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Maternal and Delivery Characteristics and Self-Reported Perceived Control During Labor. Obstet Gynecol. 2023 Jul 1;142(1):117-124. doi: 10.1097/AOG.0000000000005230. PMID 37290106
- [Derived] Costantine MM, Sandoval GJ, Grobman WA, Reddy UM, Tita ATN, Silver RM, El-Sayed YY, Wapner RJ, Rouse DJ, Saade GR, Thorp JM Jr, Chauhan SP, Chien EK, Casey BM, Srinivas SK, Swamy GK, Simhan HN; for the Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. Association of Body Mass Index With the Use of Health Care Resources in Low-Risk Nulliparous Pregnancies After 39 Weeks of Gestation. Obstet Gynecol. 2022 May 1;139(5):866-876. doi: 10.1097/AOG.0000000000004753. Epub 2022 Apr 5. PMID 35576345
- [Derived] Silver RM, Rice MM, Grobman WA, Reddy UM, Tita ATN, Mallett G, Hill K, Thom EA, El-Sayed YY, Wapner RJ, Rouse DJ, Saade GR, Thorp JM Jr, Chauhan SP, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Customized Probability of Vaginal Delivery With Induction of Labor and Expectant Management in Nulliparous Women at 39 Weeks of Gestation. Obstet Gynecol. 2020 Oct;136(4):698-705. doi: 10.1097/AOG.0000000000004046. PMID 32925634
- [Derived] Mallett G, Hill K, de Voest J, Bousleiman SZ, Allard D, Harris S, Salazar A, Clark K, Ortiz F, Bartholomew A, Dalton W, Craig J, Bickus M; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Characteristics Associated With Consent and Reasons for Declining in a Randomized Trial in Pregnancy. Obstet Gynecol. 2020 Oct;136(4):731-737. doi: 10.1097/AOG.0000000000003998. PMID 32925629
- [Derived] El-Sayed YY, Rice MM, Grobman WA, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, Wapner RJ, Rouse DJ, Saade GR, Thorp JM Jr, Chauhan SP, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Elective Labor Induction at 39 Weeks of Gestation Compared With Expectant Management: Factors Associated With Adverse Outcomes in Low-Risk Nulliparous Women. Obstet Gynecol. 2020 Oct;136(4):692-697. doi: 10.1097/AOG.0000000000004055. PMID 32925628
- [Derived] Dude A, Fette LM, Reddy UM, Tita ATN, Silver RM, El-Sayed YY, Wapner RJ, Rouse DJ, Saade GR, Thorp JM Jr, Chauhan SP, Iams JD, Chien EK, Casey BM, Srinivas SK, Swamy GK, Simhan HN; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Maternal Sense of Control During Childbirth and Infant Feeding Method. Obstet Gynecol. 2020 Mar;135(3):583-590. doi: 10.1097/AOG.0000000000003697. PMID 32028504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50,581 low-risk nulliparous women at 34 weeks 0 days gestation to 38 weeks 6 days gestation were screened for eligibility between March 2014 and August 2017 at 41 hospitals participating in the MFMU network. Women who consented were assessed again between 38 weeks 0 days gestation and 38 weeks 6 days gestation for new indications of ineligibility.
Period: Overall Study
Arm/Group | Expectant Management | Elective Induction of Labor
Started | 3044 | 3062
Completed | 3037 | 3059
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Expectant Management | Elective Induction of Labor | Total
Number analyzed (Participants) | 3044 | 3062 | 6106
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [20 to 28] | 24 [21 to 28] | 24 [20 to 28]
Age, Customized [Count of Participants; unit: Participants]
  ≥35 years | 136 | 114 | 250
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3044 | 3062 | 6106
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1359 | 1329 | 2688
  Black | 699 | 707 | 1406
  Asian | 106 | 87 | 193
  Hispanic | 808 | 866 | 1674
  Other, unknown or more than one race | 72 | 73 | 145
Married or living with partner [Count of Participants; unit: Participants] | 1798 | 1814 | 3612
Employment status [Count of Participants; unit: Participants] — Population: Data on employment status are missing for a total of 17 women.
  Participants
    number analyzed (Participants) | 3036 | 3053 | 6089
    Employed full time | 1209 | 1226 | 2435
    Employed part time | 353 | 341 | 694
    Not employed | 1474 | 1486 | 2960
Private insurance for prenatal care [Count of Participants; unit: Participants] — Population: Data is missing for one participant.
  Participants
    number analyzed (Participants) | 3044 | 3061 | 6105
    (all) | 1335 | 1404 | 2739
History of pregnancy loss [Count of Participants; unit: Participants]
  No previous pregnancy loss | 2266 | 2364 | 4630
  Previous pregnancy loss | 778 | 698 | 1476
Length of gestation at randomization [Median (Inter-Quartile Range); unit: weeks] | 38.3 [38.0 to 38.6] | 38.3 [38.0 to 38.6] | 38.3 [38.0 to 38.6]
Method of conception [Count of Participants; unit: Participants]
  In vitro fertilization | 47 | 56 | 103
  Ovulation inducation or artificial insemination | 24 | 30 | 54
  Spontaneous | 2973 | 2976 | 5949
Smoked cigarettes [Count of Participants; unit: Participants] | 242 | 224 | 466
Drank alcohol [Count of Participants; unit: Participants] — Population: Data are missing for 1 participant
  Participants
    number analyzed (Participants) | 3043 | 3062 | 6105
    (all) | 107 | 133 | 240
BMI at randomization [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Data are missing for 30 women
  kg/m^2
    number analyzed (Participants) | 3027 | 3049 | 6076
    (all) | 30.3 [27.3 to 35.0] | 30.5 [27.3 to 34.6] | 30.4 [27.3 to 34.8]
BMI ≥30 at randomization [Count of Participants; unit: Participants] — Participants who had a body-mass index (BMI) of greater than or equal to 30 at randomization. BMI is weight in kilograms divided by the square of the height in meters. Population: Data are missing for 30 women
  Participants
    number analyzed (Participants) | 3027 | 3049 | 6076
    (all) | 1575 | 1632 | 3207
Modified Bishop Score at randomization [Median (Inter-Quartile Range); unit: units on a scale] — Modified Bishop scores range from 0 to 12, with lower scores associated with a higher chance of cesarean delivery. Population: Data is missing for 2 participants.
  units on a scale
    number analyzed (Participants) | 3042 | 3062 | 6104
    (all) | 4 [2 to 5] | 4 [2 to 5] | 4 [2 to 5]
Modified Bishop score <5 at randomization [Count of Participants; unit: Participants] — Modified Bishop scores range from 0 to 12, with lower scores associated with a higher chance of cesarean delivery Population: Data is missing for 2 participants
  Participants
    number analyzed (Participants) | 3042 | 3062 | 6104
    (all) | 1954 | 1919 | 3873

OUTCOME MEASURES:

1. Primary Outcome: Composite of Severe Neonatal Morbidity and Perinatal Mortality
Description: Includes any one of:
  * Perinatal death
  * Need for respiratory support within 72 hours after birth
  * Apgar score of 3 or less at 5 minutes
  * Hypoxic-ischemic encephalopathy
  * Seizure
  * Infection (confirmed sepsis or pneumonia)
  * Meconium aspiration system
  * Birth trauma (bone fracture, neurologic injury or retinal hemorrhage)
  * Intracranial or subaleal hemorrhage
  * Hypotension requiring vasopressor support
Time Frame: delivery through 72 hours after birth
Population: The analysis was intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 164 | 132
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.049, Chi-squared; Group sequential method to control type I error w/ Lan-DeMets characterization of O'Brien-Fleming boundary. 2-tailed p-value <0.46 considered stat sig; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.64 to 1.00] — One interim analysis was performed; in final analysis of the primary outcome, a two-tailed P value of less than 0.046 considered to indicate statistical significance. Since adjustment is minimal, we report 95% confidence interval for relative risk

2. Primary Outcome: Perinatal Death (Component of Primary Outcome)
Description: Perinatal death includes antepartum stillbirth, intrapartum stillbirth and neonatal death
Time Frame: antepartum pregnancy period through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 3 | 2
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.12 to 3.33] — Exact confidence intervals are provided for rare outcomes. Widths of the confidence intervals for components of the primary outcome have not been adjusted for multiplicity, and should not be used to infer definitive effects of management strategies

3. Primary Outcome: Number of Participant Infants Requiring Respiratory Support (Component of Primary Outcome)
Description: Respiratory support includes mechanical ventilation, continuous positive airway pressure or high flow nasal cannula and cardiorespiratory resuscitation
Time Frame: Delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 127 | 91
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.55 to 0.93]

4. Primary Outcome: Number of Infants With Apgar Score ≤3 at 5 Minutes (Component of Primary Outcome)
Description: The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: Delivery through 5 minutes after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 18 | 12
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.32 to 1.37] — Widths of the confidence intervals for components of the primary outcome have not been adjusted for multiplicity, and should not be used to infer definitive effects of management strategies

5. Primary Outcome: Number of Infants With Neonatal Hypoxic-ischemic Encelphalopathy (Component of Primary Outcome)
Time Frame: delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 20 | 14
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.35 to 1.37] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: Number of Infants With Neonatal Seizure (Component of Primary Outcome)
Time Frame: Delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 4 | 11
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 2.74, 95% CI 2-sided [0.91 to 8.12] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Number of Infants With Neonatal Infection (Component of Primary Outcome)
Description: Neonatal infection includes confirmed sepsis and/or confirmed pneumonia
Time Frame: delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 12 | 9
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.31 to 1.76] — [estimate comment as in outcome 4, analysis 1]

8. Primary Outcome: Number of Infants With Meconium Aspiration Syndrome (Component of Primary Outcome)
Time Frame: Delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 26 | 17
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.35 to 1.19] — [estimate comment as in outcome 4, analysis 1]

9. Primary Outcome: Number of Infants With Birth Trauma (Component of Primary Outcome)
Description: Birth trauma includes clavicular, skull or other fracture; brachial plexus palsy, facial nerve palsy, retinal hemorrhage or vocal cord paralysis
Time Frame: During the Delivery process
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 18 | 14
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.38 to 1.55] — [estimate comment as in outcome 4, analysis 1]

10. Primary Outcome: Number of Infants With Intracranial or Subgaleal Hemorrhage (Component of Primary Outcome)
Description: Intracranial or subgaleal hemorrhage includes Intraventricular hemorrhage grades III or IV, subdural hematoma, subarachnoid hematoma, and subgaleal hematoma
Time Frame: delivery through disharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 7 | 9
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.48 to 3.42] — [estimate comment as in outcome 4, analysis 1]

11. Primary Outcome: Hypotension Requiring Vasopressor Support (Component of Primary Outcome)
Time Frame: delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 5 | 2
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; Risk Ratio (RR) = 0.40, 95% CI 2-sided [0.06 to 1.79] — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Number of Participants With Cesarean Delivery
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 674 | 569
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p < 0.001, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.76 to 0.93]

13. Secondary Outcome: Number of Participants Who Had Uterine Incisional Extension at Cesarean Delivery
Description: Incisional extensions at cesarean section, including J shape or T shape; or cervical traumas
Time Frame: delivery
Population: Neonatal length of hospital stay missing in 5 (2 induction group (IOL); 3 expectant-management group (EM)); incisional extensions at cesarean section missing in 9 (5 IOL; 4 EM); breastfeeding status at 4-8 wk after delivery missing in 642 (299 IOL; 343 EM).
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 48 | 28
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.02, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.36 to 0.92]

14. Secondary Outcome: Participants Who Had Operative Vaginal Delivery
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 258 | 222
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.07, Chi-squared; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.72 to 1.01]

15. Secondary Outcome: Number of Participants Who Had Chorioamnionitis
Description: Chorioamnionitis, defined as a clinical diagnosis before delivery
Time Frame: at any time from randomization through delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 429 | 407
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.35, Chi-squared; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.83 to 1.07]

16. Secondary Outcome: Number of Participants With Third or Fourth Degree Perineal Laceration
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 89 | 103
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.33, Chi-squared; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.87 to 1.52]

17. Secondary Outcome: Number of Maternal Deaths
Description: Maternal death at anytime between randomization and hospital discharge.
Time Frame: from randomization to hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 0 | 0

18. Secondary Outcome: Number of Participants Admitted to Intensive Care Unit (ICU)
Description: Admission of the participant to the intensive care unit (ICU)
Time Frame: delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 8 | 4
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.26, Chi-squared; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.13 to 1.55] — Exact confidence intervals are provided for rare outcomes

19. Secondary Outcome: Number of Participants Experiencing Hypertensive Disorder of Pregnancy
Time Frame: Randomization to hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 427 | 277
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p < 0.001, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.56 to 0.74]

20. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Description: defined as any of the following:
  * Transfusion
  * Non-elective hysterectomy
  * Use of two or more uterotonics other than oxytocin
  * Other surgical interventions such as uterine compression sutures, uterine artery ligation, embolization, hypogastric ligation, or balloon tamponade
  * Curettage
Time Frame: delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 137 | 142
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.81, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.82 to 1.29]

21. Secondary Outcome: Labor Agentry Scale Scores
Description: Scores on the Labor Agentry Scale range from 29 to 203, with higher scores indicating greater perceived control during childbirth; included are women who had spontaneous labor, labor that started spontaneously but then was augmented, or induced labor.
Time Frame: Between 6 hours after delivery and 8 weeks after delivery
Population: Data for 6 to 96 hours after delivery are missing for 288 women (127 in the induction group and 161 in the expectant-management group); data for 4 to 8 weeks after delivery are missing for 736 women (349 in the induction group and 387 in the expectant-management group).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
score on a scale
  At 6-96 hr after delivery: number analyzed (Participants) | 2876 | 2932
  At 6-96 hr after delivery | 164 [143 to 181] | 168 [148 to 183]
  At 4-8 weeks after delivery: number analyzed (Participants) | 2650 | 2710
  At 4-8 weeks after delivery | 174 [154 to 188] | 176 [157 to 189]
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Analysis for 6-96 hours after delivery; Test type: Superiority; p < 0.001, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method
Statistical Analysis 2: Comparison: Expectant Management vs Elective Induction of Labor; Analysis for 4-8 weeks after delivery; Test type: Superiority; p = 0.01, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method

22. Secondary Outcome: Labor Pain Scores
Description: Labor pain was scored according to a 10-point Likert scale, with higher scores indicating greater pain; included are women who had spontaneous labor, labor that started spontaneously but then was augmented, or induced labor.
Time Frame: During labor and delivery
Population: Data on worst score are missing for 274 women (110 in the induction group and 164 in the expectant-management group); data on overall score are missing for 275 women (110 in the induction group and 165 in the expectant-management group).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
score on a scale
  Worst score: number analyzed (Participants) | 2873 | 2949
  Worst score | 9 [8 to 10] | 8 [7 to 10]
  Overall score: number analyzed (Participants) | 2872 | 2949
  Overall score | 7 [5 to 9] | 7 [5 to 8]
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Analysis for Worst labor pain score; Test type: Superiority; p < 0.001, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method
Statistical Analysis 2: Comparison: Expectant Management vs Elective Induction of Labor; Analysis for Overall labor pain score; Test type: Superiority; p < 0.001, Chi-squared — The P value remained significant after controlling for multiple comparisons with the false discovery rate method

23. Secondary Outcome: Number of Participants With Maternal Postpartum Infection
Description: Defined as any of the following:
  * Clinical diagnosis of endometritis
  * Wound reopened for hematoma, seroma, infection or other reasons
  * Cellulitis requiring antibiotics
  * Pneumonia
  * Pyelonephritis
  * Bacteremia - unknown source
  * Septic pelvic thrombosis
Time Frame: delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 65 | 50
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.15, Chi-squared; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.53 to 1.10]

24. Secondary Outcome: Number of Participants With Venous Thromboembolism
Description: Maternal deep venous thrombosis or pulmonary embolism
Time Frame: delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 1 | 2
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 1.00, Chi-squared; The P-values has not been adjusted for multiplicity of comparisons of secondary outcomes; Risk Ratio (RR) = 1.99, 95% CI 2-sided [0.26 to 26.8] — Exact confidence intervals are provided for rare outcomes

25. Secondary Outcome: Number of Participants With Indications for Cesarean Delivery
Description: Number of participants with indications for cesarean delivery including dystocia, non-reassuring fetal status or other indication
Time Frame: Labor and delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants
  Dystocia | 289 | 259
  Non-reassuring fetal status | 332 | 275
  Other c-section indication | 53 | 35

26. Secondary Outcome: Duration of Respiratory Support
Description: including ventilator, CPAP, high-flow nasal cannula (HFNC)
Time Frame: delivery through hospital discharge
Population: One neonate had cardiorespiratory resuscitation and 0 days on mechanical ventilation, continuous positive airway pressure or high flow nasal cannula.
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants
  0 days | 2911 | 2968
  1 day | 70 | 55
  Greater than 1 day | 56 | 36
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.01, Cochran-Armitage trend test

27. Secondary Outcome: Number of Infants With Cephalohematoma
Time Frame: delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 90 | 83
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.56, Chi-squared; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.68 to 1.23]

28. Secondary Outcome: Shoulder Dystocia
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 65 | 59
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.56, Chi-squared; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.64 to 1.28]

29. Secondary Outcome: Number of Infants Who Had Transfusion of Blood Products or Blood
Time Frame: delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 5 | 4
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.75, Chi-squared; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.20 to 2.74] — Exact confidence intervals are provided for rare outcomes

30. Secondary Outcome: Number of Infants With Hyperbilirubinemia
Description: Hyperbilirubinemia requiring phototherapy or exchange transfusion
Time Frame: delivery through discharge
Population: Data were missing for 4 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3034 | 3058
Participants | 142 | 145
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.91, Chi-squared; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.81 to 1.27]

31. Secondary Outcome: Number of Infants With Neonatal Hypoglycemia
Description: glucose < 35 mg/dl and requiring IV therapy
Time Frame: delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 35 | 37
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.84, Chi-squared; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.66 to 1.66]

32. Secondary Outcome: Number Infants Admitted to NICU or Intermediate Care
Description: Number infants admitted to intensive care unit (NICU) or intermediate care unit
Time Frame: delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants | 394 | 358
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.13, Chi-squared; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.79 to 1.03]

33. Secondary Outcome: Number of Hours on the Labor and Delivery Unit
Description: Median duration of stay in labor and delivery unit
Time Frame: Hours from admission to L&D to discharge from L&D
Population: Excludes 7 women who delivered before admission to the labor and delivery unit. Data are missing for 2 women.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3036 | 3058
hours | 14 [9 to 20] | 20 [13 to 28]
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p < 0.001, Wilcoxon Rank-Sum

34. Secondary Outcome: Maternal Postpartum Length of Hospital Stay
Time Frame: delivery through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants
  <2 days | 317 | 322
  2 days | 2084 | 2191
  3 days | 452 | 399
  4 days | 166 | 130
  >4 days | 18 | 17
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.01, Cochran-Armitage trend test — The P value remained significant after controlling for multiple comparisons with the false discovery rate method

35. Secondary Outcome: Neonatal Length of Hospital Stay
Time Frame: delivery through hospital discharge
Population: Data is missing for 5 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3034 | 3057
Participants
  <2 days | 315 | 321
  2 days | 1904 | 2030
  3 days | 498 | 457
  4 days | 189 | 142
  >4 days | 128 | 107
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Test type: Superiority; p = 0.002, Cochran-Armitage trend test — The P value remained significant after controlling for multiple comparisons with the false discovery rate method

36. Secondary Outcome: Number of Participants With Indications for Operative Vaginal Delivery
Description: Number of participants with indications for operative vaginal delivery including dystocia, non-reassuring fetal status and other indications
Time Frame: Labor and delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants
  Dystocia | 94 | 101
  Non-reassuring fetal status | 156 | 119
  Other indication | 6 | 1

37. Secondary Outcome: Number of Participants and Breastfeeding Status at 4-8 Weeks After Delivery
Description: Breastfeeding status includes breastfeeding, breastfeeding and formula feeding, or formula feeding
Time Frame: 4-8 weeks after delivery
Population: breastfeeding status at 4-8 wk after delivery missing in 642 (299 IOL; 343 EM)
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Elective Induction of Labor
Number analyzed (Participants) | 3037 | 3059
Participants
  Breastfeeding: number analyzed (Participants) | 2694 | 2760
  Breastfeeding | 891 | 916
  Breast Feeding and Formula Feeding: number analyzed (Participants) | 2694 | 2760
  Breast Feeding and Formula Feeding | 831 | 863
  Formula Feeding: number analyzed (Participants) | 2694 | 2760
  Formula Feeding | 972 | 981
Statistical Analysis 1: Comparison: Expectant Management vs Elective Induction of Labor; Multinomial logistic regression using participants who are breastfeeding only as the reference group. This analysis compares the participants who are breastfeeding and formula feeding to participants who are only breastfeeding; Test type: Other; p = 0.88, Regression, Logistic — Odds ratios from multinomial logistic regression; Odds Ratio, log = 1.01, 95% CI 2-sided [0.89 to 1.15]
Statistical Analysis 2: Comparison: Expectant Management vs Elective Induction of Labor; Multinomial logistic regression using participants who are breastfeeding only as the reference group. This analysis compares the participants who are only formula feeding to participants who are only breastfeeding; Test type: Other; p = 0.78, Regression, Logistic; Odds Ratio, log = 0.98, 95% CI 2-sided [0.86 to 1.12]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected and evaluated from the date of randomization (between 38 weeks, 0 days gestation and 38 weeks, 6 days gestation) through approximately 8 weeks postpartum. This time frame encompasses between 9 and 12 weeks.
Description: The primary and secondary outcomes comprise all the adverse events that occurred. We expect this is different than, for example, a medication trial in which adverse events other than those related to the outcomes may occur.
Arm/Group | Expectant Management | Elective Induction of Labor
All-Cause Mortality (participants affected / at risk) | 3/3059 | 2/3037
Serious Adverse Events (participants affected / at risk) | 3/3037 | 2/3059
Other Adverse Events (participants affected / at risk) | 0/3037 | 0/3059
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expectant Management (N=3037) | Elective Induction of Labor (N=3059)
Perinatal Death (Pregnancy, puerperium and perinatal conditions) | 3 (3037) | 2 (3059)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-10-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT01990612/Prot_SAP_ICF_000.pdf